CLINICAL TRIAL: NCT00704990
Title: The Safety and Efficacy of a Compound Natural Health Product in Children With Attention Deficit/Hyperactivity Disorder: A Pilot Study
Brief Title: Combination Natural Health Product in Children With Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kieran Cooley (Other)
Collaborators: The Canadian College of Naturopathic Medicine (Other); University of Toronto (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor-Investigator, Kieran Cooley, Principle Investigator, The Canadian College of Naturopathic Medicine
Organization: The Canadian College of Naturopathic Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCNM-083-ADHD
Record Dates: First submitted 2008-06-20; First posted 2008-06-25 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Disorder; Pediatrics; Attention; Impulsivity; Complementary Therapies
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Impulsive Behavior | interventions — Zinc; Magnesium; Vitamin B 6; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): All study participants take part in the experimental arm
  Interventions: Dietary Supplement: Zinc, Magnesium, Vitamin B6, Vitamin C (Compound Natural Health Product for ADHD)

INTERVENTIONS:
Dietary Supplement: Zinc, Magnesium, Vitamin B6, Vitamin C (Compound Natural Health Product for ADHD) — Weight based dosing of a chewable natural health product containing 15-35 mg zinc citrate, 150-350 mg magnesium lactate, 30-70 mg pyridoxine hydrochloride and 150-350 mg calcium ascorbate. Participants will take weight based dose two times during the day with meals for a 10 week period
  Other Names: Zinc; Magnesium; Vitamin B6; Vitamin C

SUMMARY:
Attention deficit/hyperactivity disorder (ADHD) is a chronic neurobehavioural disorder often diagnosed in childhood years. Complementary/alternative treatments including natural health products (NHPs) are used by children with ADHD despite limited information on their safety or usefulness. Some evidence suggests children with ADHD have a greater need for zinc, magnesium, vitamin B6 and vitamin C. This study will supplement a small number of children diagnosed with ADHD with therapeutic levels of these nutrients over 10 weeks to get a better understanding of the safety and possible benefit of using these nutrients to treat symptoms associated with ADHD.

DETAILED DESCRIPTION:
The is an open-label study. Children diagnosed with ADHD will be provided with a weight-based dose of a chewable natural health product containing zinc, magnesium, vitamin B6 and vitamin C for 10 weeks with an additional follow-up post intervention at 20 weeks. Severity of ADHD symptoms will be measured at baseline, week 5 and week 10 using the Connor-3 Parent and SNAP-IV validated questionnaires. Nutritional status will be monitored at baseline and week 10 for changes in serum zinc and erythrocyte magnesium. Children will be monitored for any adverse reactions that may occur using the investigational product.Following the informed consent process, participants will undergo a structured psychiatric interview prior to enrollment and will have 4 30 minute study visits and 2 10 minute telephone calls throughout the study. Blood samples will be taken 2 times with the use of a topical anesthetic to decrease sensation during the blood draw. Once enrolled, children can withdraw from the study at any time if assent to participate is withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children age 6-12 diagnosed with ADHD of any subtype according to DSM-IV criteria. A structured diagnostic interview (Kiddie Sads Present and Lifetime Version) will be conducted to confirm diagnosis of ADHD and assess for comorbid mental health disorders.
* Primary caregiver (parent or guardian) has given informed consent; child participant gives ongoing assent throughout the study.

Exclusion Criteria:

* Changes to participants' ADHD medication within 6 weeks of study onset.
* Diagnosis of additional mental health disorder using the Kiddie Sads.
* Diagnosis of cancer.
* Antibiotic use for periods greater than 2 weeks within the 10 weeks prior to the study
* Diagnosis of Type 1 diabetes and insulin use
* Low serum ferritin/iron deficiency (<30 ng/ml)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Connors-3 Parent Rating Scale | Baseline, week 5, week 10 and follow-up at week 20

SECONDARY OUTCOMES:
Nutritional status of zinc and magnesium | Week 0 and week 10
Adverse events | Throughout study
SNAP-IV Parent ADHD questionnaire | Week 0, week 5 and week 10

CONTACTS AND LOCATIONS:
Overall Officials: Heather Boon, PhD, Principal Investigator — University of Toronto; Umesh Jain, MD, Study Director — The Center for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Robert Schad Naturopathic Clinic, Toronto, Ontario
  - The Center for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- See also: Abstract of results presented at the American Association of Naturopathic Physician's convention in August, 2010 — http://naturalmedicinejournal.net/pdf/NMJ_SEP10_ABS.pdf